CLINICAL TRIAL: NCT02476656
Title: Placental Inflammation in Prenatal Care
Acronym: PINC
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Other Study IDs: Pro#00037264
Record Dates: First submitted 2015-05-19; First posted 2015-06-19 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2016-10

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GPNC: CenteringPregnancy group prenatal care
- IPNC: Individual prenatal care

SUMMARY:
Objective of study is to explore expression of stress-related genes and inflammation in placentas and umbilical cord blood for women participating in group prenatal care compared with women receiving individual prenatal care.

DETAILED DESCRIPTION:
This study aims to evaluate levels of inflammatory markers and genetic indicators of stress an inflammation in the placentas and umbilical cord blood in pregnancies that undergo group prenatal care as compared to traditional prenatal care. The investigators know that women receiving group prenatal care have fewer spontaneous preterm deliveries. What is not known is the mechanism behind this difference. By collecting umbilical cord blood samples and placentas of 40 women at the time of delivery, the investigators hope to study expression of stress-related genes and levels of inflammatory markers at the maternal-fetal interface.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Singleton pregnancy

Exclusion Criteria:

* Presence of known fetal congenital anomalies (lethal anomaly or anomalies that may lead to early delivery or increased risk of neonatal death).
* Presence of known chromosomal abnormalities
* Progesterone treatment during the current pregnancy after 14 weeks
* Chronic corticosteroid (i.e. Prednisone or other steroids) treatment during the current pregnancy (not including inhalers or topical)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: preganant women who present for delivery at term at Greenville Health System with the Obstetrics Teaching Service
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers (CRP, IL-6) of cord blood | drawn from the umbilical cord within 15 minutes of delivery
  Circulating concentrations of C-reactive protein and interleukin-6 will be quantified in serum harvested from umblical blood

SECONDARY OUTCOMES:
Genome wide expression profiling of cord blood | drawn from the umbilical cord within 15 minutes of delivery
  Mononuclear cells will be isolated from umbilical blood using density gradient centrifugation. RNA will be extracted using Qiagen RNeasy Mini Kits, and quality/quantity checks performed using an Agilent NanoDrop BioAnalyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Picklesimer, MD, MSPH, Principal Investigator — Prisma Health-Upstate